CLINICAL TRIAL: NCT00467090
Title: Expanding the Phenotype of the LRRK-2 Mutation in Individuals With History of Parkinson s Disease and Their Relatives: a Prospective Study
Brief Title: Characteristics of Parkinson s Disease Associated With the LRRK-2 Gene Mutation
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070137; 07-N-0137
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-02-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Gene; Genetic; Family Studies; LRRK-2; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will identify symptoms and other characteristics of Parkinson s disease that may be associated with changes in a gene called leucine-rich repeat kinase 2 (LRRK2). Changes in this gene have been found in patients with and without a family history of Parkinson s disease. This study will examine people with Parkinson s disease to try to identify how symptoms develop over time. First-degree relatives of patients will also be studied.

People 18 years of age or older with Parkinson s disease or people who have a first-degree relative with Parkinson s disease may be eligible for this study.

Participants visit the NIH Clinical Center every other year for 10 years for some or all of the procedures listed below. Each visit requires 3-4 days of testing, which may be done on an inpatient or outpatient basis. Telephone interviews are conducted during the alternate years.

* History and physical examination.
* Smell testing: Subjects are asked to identify 40 different scents.
* Sensory testing: Objects with grooves and ridges are touched to subjects fingertips. With their eyes closed, the subjects are asked to say which way the grooves and ridges run on the objects.
* Neuropsychological evaluation: Subjects are asked about their memory and thinking and may be asked to complete some pen and paper tests.
* Psychiatric evaluation: Subjects are asked about psychiatric symptoms, including anxiety and depression.
* Blood drawing: Blood is drawn through a needle in the arm.
* Magnetic imaging resonance (MRI) scans of the brain: MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. During the test, subjects lie on a table that can slide in and out of the MRI scanner (a metal cylinder surrounded by a strong magnetic field). The procedure lasts about 30 minutes, during which the subjects may be asked to lie still for up to 5 minutes at a time.
* Transcranial sonography (TCS): TCS uses sound waves to obtain images of the brain. Subjects lie on their back and an ultrasound device is moved around the scalp.
* Sleep study (1-2 night hospital admission): Subjects brain waves are recorded during sleep using electroencephalography (EEG). Their breathing rate, pulse and oxygen level are also monitored.
* Questionnaire: Subjects complete several questionnaires designed to obtain information on symptoms or traits that have been reported to be associated with Parkinson s disease.

DETAILED DESCRIPTION:
Parkinson s disease is a common neurological condition that was originally thought to develop from environmental factors. More recently, genetic factors have been implicated. In this study, we are interested in studying the phenotypic presentation of patients with Parkinson s disease due to a specific defect in a gene called the Leucine rich repeat kinase 2 gene (LRRK2) found in some patients with Parkinson s disease. In addition, we plan to study family members whose genetic status is unknown to develop a pre-clinical description of Parkinson s disease progression.

OBJECTIVE:

1. To develop a pre-clinical description in first-degree family members of patients with Parkinson s disease who have the LRRK2 mutation. The first-degree relative may or may not carry the LRRK2 mutation.
2. To phenotypically characterize Parkinson s disease patients who have the LRRK2 mutation.

STUDY POPULATION:

200 adult subjects including:

1. Patients with a diagnosis of PD due to LRRK2 mutation
2. First degree family members of patients with PD who have the LRRK2 mutation.

DESIGN:

This will be a longitudinal prospective natural history study.

OUTCOME MEASURES:

1. Pre-clinical signs of disease in first degree relatives of Parkinson s disease patients who have the LRRK2 mutation.
2. Characterization of a pre-clinical phenotype in first degree relatives of LRRK2 positive Parkinson s disease patients.
3. Progression of Parkinson s disease patients who have the LRRK2 mutation.
4. Genotypic characterization of first-degree relatives
5. RNA expression profile determination comparing mutation carriers to non-mutation carriers in search for early biomarkers

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects at least 18 years of age.
  2. Ability to provide consent or have appointed a Durable Power of Attorney able to provide consent.
  3. Patients with a diagnosis of PD with a known LRRK2 mutation.

     OR
  4. First degree relatives without a diagnosis of PD with a family history suggestive of inherited PD due to LRRK2 mutations.

EXCLUSION CRITERIA:

1. Subjects with a history of severe head injury, encephalitis, chronic use of drugs that cause parkinsonism or a clinical history of strokes.
2. For the magnetic resonance imaging (MRI), exclusion criteria include the following: pregnancy, pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments. Patients will be screened for these conditions prior to having the MRI scan performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-04-23; Study Completion 2014-02-03

CONTACTS AND LOCATIONS:
Overall Officials: Grisel J Lopez, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Braak H, Braak E. Pathoanatomy of Parkinson's disease. J Neurol. 2000 Apr;247 Suppl 2:II3-10. doi: 10.1007/PL00007758. PMID 10991663
- [Background] Nussbaum RL, Ellis CE. Alzheimer's disease and Parkinson's disease. N Engl J Med. 2003 Apr 3;348(14):1356-64. doi: 10.1056/NEJM2003ra020003. No abstract available. PMID 12672864
- [Background] Litvan I, Bhatia KP, Burn DJ, Goetz CG, Lang AE, McKeith I, Quinn N, Sethi KD, Shults C, Wenning GK; Movement Disorders Society Scientific Issues Committee. Movement Disorders Society Scientific Issues Committee report: SIC Task Force appraisal of clinical diagnostic criteria for Parkinsonian disorders. Mov Disord. 2003 May;18(5):467-86. doi: 10.1002/mds.10459. PMID 12722160